CLINICAL TRIAL: NCT02666274
Title: Feasibility Studies to Inform Novel Proposals to Avert Community-Based Antimicrobial Resistance Spread
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: RJ115/N354
Record Dates: First submitted 2016-01-18; First posted 2016-01-28 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: Gram-Negative Bacterial Infections
Keywords: carbapenem resistance; bacterial carriage; multi-drug resistant gram negative bacteria
MeSH Terms: conditions — Gram-Negative Bacterial Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — stool samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- RK Group: participants colonised with Klebsiella spp. resistant to either 3GC or carbapenems (RK cohort of index carriers of Resistant Klebsiella)

SUMMARY:
There are many bacteria that naturally live in our gut and are essential for good health. These bacteria have a variety of helpful functions, such as aiding digestion, synthesizing vitamins, repressing the growth of harmful bacteria and defending against some diseases. The desirable bacteria that live in the gut are collectively known as 'gut flora', or more appropriately, as 'gut microbiota'.

The less desirable resistant bacteria, however, can also be carried in a person's gut for prolonged periods of time and be found in the stools without causing illness. Persons that carry the resistant bacteria in the gut are known as "carriers" and they require no treatment. Knowing that a person carries resistant bacteria is helpful, because it will inform the choice of antibiotic if the person were to become unwell or had an intervention such as surgery in the future.

There is some evidence that resistant bacteria found in the stools can sometimes be passed from one person to another and eventually make someone ill if they infect (invade) their body. The investigators do not know how often this may happen, or how much carrying resistant bacteria in the stools may facilitate the spread of resistant bacteria in the population. It is important to address these questions and study ways to stop the resistant bacteria from spreading to safeguard the efficacy of antibiotics.

DETAILED DESCRIPTION:
1. Study A. Mapping of resistant gram negative bacteria (RGNB) in the community: Based on RGNB clinical isolates as a proxy for gut colonising RGNB and residential Lower Layer Super Output Area (LSOA) data retrieved from laboratory information systems of a hospital cohort, to describe the geographical distribution of RGNB in South East London in relation to demographic, cultural and socioeconomic indicators and to investigate whether geographical clustering of resistance, compatible with the occurrence of community based transmission hotspots, occurs in our local community.
2. Study B. Tracking gut colonisation with carbapenem resistant Klebsiella spp. or Klebsiella spp. resistant to third generation cephalosporins (3GC), herein referred to as 'Resistant Klebsiella' (RK):

To investigate the duration of gut colonisation with Klebsiella spp. in a small cohort of discharged hospital patients with resistance to the carbapenems (eg. meropenem), defined by presence of either blaKPC, blaNDM, blaIMP , blaVIM or blaOXA48 genes, or Klebsiella spp. with resistance to the 3GC (eg. ceftazidime), defined by presence of blaCTX_M or AmpC βlactamase genes. To determine the occurrence of participant to participant RK transmission events within a household, in relation to gut bacterial load and the gut microbiota profile. To characterise over time, the gut microbiota profile of participants colonised with RK as compared to participants who only carry antibiotic susceptible enterobacteria in the gut. It is beyond the scope of our feasibility study to enrol a sample of persons that is representative of the wider population, or to account for sample size and power calculations that would allow for characterisation of statistically meaningful associations.

ELIGIBILITY:
Inclusion Criteria:

* Study A ('Mapping'): Retrospective data collection from the hospital laboratory information system on patients diagnosed with infection and/or colonisation by relevant gram negative bacteria and antibiotic resistance profile.
* Study B ('Tracking'):

  * Inclusion criteria for index participants are being at least 16 years of age, able to consent for themselves and to communicate in English at the time of being invited to participate in the study. Inclusion criteria for index participants in the RK group include gut colonisation by Klebsiella spp. with resistance to carbapenems or third generation cephalosporins, as demonstrated by the analysis of a stool sample provided at baseline. Inclusion criteria for index participants in the control group, are lack of colonisation by bacteria resistant to third generation cephalosporins or carbapenems, as demonstrated by the analysis of a stool sample provided at baseline and at 6 months after discharge from hospital.
  * Inclusion criteria for network participants are persons of any age who are sharing the household with an index participant in the RK group and who meet the definition of usual household resident.

Exclusion Criteria:

* Study A ('Mapping'): Exclusion criteria include data from penitentiary patients.

Study B ('Tracking'):

* Exclusion criteria for index participants are those not meeting the inclusion criteria, penitentiary patients, those with no fixed adobe or not residing in a household space as defined in this study, and those living alone.
* Exclusion criteria for network participants are those not meeting the inclusion criteria, those meeting exclusion criteria as defined for index participants, those who are adults unable to consent for themselves, and those who are not able to communicate in English.
* Exclusion criteria for households are those not meeting the inclusion criteria, those where the index participant resides alone (i.e. no other usual residents in the household), those were at least one resident is not eligible for inclusion (including where a resident does not meet the definition of usual resident), those where at least one usual resident does not want to take part in the study, and those which are more than one hour commute from the study site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any adult hospitalized patient at Guy's and St Thomas' Foundation Trust who carries resistant gram negative bacteria on a screening or clinical sample
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2015-12; Primary Completion 2017-01 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Transmission of resistant gram negative bacteria from index participants and network participants | 6 months
  To measure household transmission between index participants and household members of resistant bacteria through collection of stool samples.
Length of Gut Carriage of resistant gram negative bacteria in index participants | 6 months
  Measure how long resistant gram negative bacteria persist in the stool by measuring carriage of bacteria in longitudinal stool samples

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Edgeworth, MBBS, Principal Investigator — Guy's and St Thomas NHS Foundation Trust
Locations (1):
- Guy's and St Thomas' NHS Foundation Trust, London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No